CLINICAL TRIAL: NCT03809871
Title: Biomarker Feedback on Health and Wellbeing and Exercise Adherence Following a 6 Month Weight Management Course: A Pilot Study
Brief Title: Biomarker Feedback on Health and Wellbeing and Exercise Adherence Following a 6 Month Weight Management Course
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hertfordshire (Other)
Collaborators: Medichecks (Unknown); Watford FC Community Sports and Education Trust (Unknown)
Responsible Party: Principal Investigator, Lindsay Bottoms, Research Lead for Sport, Health and Exercise, University of Hertfordshire
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LMS
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Exercise Training; Biomarkers
Keywords: exercise training; weight management; biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biomarker group (Experimental): These participants will receive information about cardiometabolic biomarkers pre and post weight management course
  Interventions: Biological: Cardiometabolic biomarkers
- Control group (No Intervention): They will receive the same weight management programme as the experimental group, but they will not have biomarker information.

INTERVENTIONS:
Biological: Cardiometabolic biomarkers — This is for measures of cholesterol (HDL, LDL and total cholesterol), blood glucose and HbA1c, vitamin D, vitamin B12 and iron levels.
  Arms: Biomarker group

SUMMARY:
Participants who have signed up to the Watford Football Club Community and Education Trust Weight management programme called Shape Up will be approached to see if they would like to take part in this research study. Their participation in the Shape Up programme will not be affected if they do not choose to opt in to the research component. Fifty participants will be recruited and randomised in to one of two groups. One group will be the control group and they will undertake the Shape Up programme as normal and will be asked to complete some questionnaires in week 1, week 12 and then at 12 weeks follow up. The intervention group will be asked to complete the same questionnaires and will also have a venous blood sample taken at week 1, 12 and then at 12 weeks follow up. This is for measures of cholesterol, sugar, vitamin D, vitamin B12 and iron. The participants will receive a report from a medical doctor in layman terms on these results a week later and will have access to their data on an online portal set up by Medichecks.

The weight management programme is based on a behaviour change programme where the participants attend a 90-minute session for 12 weeks, and they are then supported for another 12 weeks following the end of the supervision. The participants have weight and BMI measured at week 1, 12 and 12 weeks follow up. Each session consists of an education component followed by an exercise component. Initially, the education part is longer and the exercise is shorter, but as the programme progresses the education part becomes shorter and the exercise longer. The education programme includes topics such as healthy eating, increased physical activity and stress. The exercise programme includes whole body activities such as circuit training as well as other group exercise such as football.

The questionnaires will include The Treatment Self-Regulation Questionnaire which will identify the motivation behind the participants' health. A general health questionnaire which is a subjective measure of health (Euro qol EQ-5). The Mental Component Summary of the 12- item Short Form (SF12) which measures emotional quality of life. Physical activity will be measured through the short Active Lives Questionnaire. All these questionnaires have been attached as appendices.

All participants will complete an exit telephone interview from the study to determine qualitative feedback on their experience of the study and to explore whether the biomarkers influenced their motivation to change their lifestyle. Some example questions have been attached.

This is just a feasibility study, therefore no hypothesis testing will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* BMI >28
* No injuries

Exclusion Criteria:

* Injury preventing from participating in exercise
* fear of needles
* does not pass a physical activity readiness questionnaire

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Behaviour regulation | 12 months
  To determine the behaviour regulation by measuring autonmoic regulation versus controlled regulation through the use of the Treatment Self-Regulation Questionnaire.
  An average of the scores on the subscale for autoregulation and also for the controlled regulation questions will be calculated. Scores will be from 1-7 for both sub scales.
Subjective health measure | 12 months
  A standardised measure of health status will be calculated using the Euro qol EQ-5 questionnaire. There are 5 dimensions to the questionnaire (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and each is rated from 1-5. An average of the 5 is calculated as a general health score. A visual analogue scale is also presented for a self related health measure and this is from 0-100. 100 being the best health you can imagine and 0 being the worst health you can imagine.
Physical Activity | 12 months
  Amount of physical activity measured through the short Active Lives questionnaire. The amount of minutes where breathing is increased will be calculated per week.
  For each activity that respondents indicate was sufficient to raise their breathing rate, the total number of days is multiplied by the usual minutes spent undertaking the activity to give a measure of total minutes over the 7-day period for that activity.
  The respondent's final score is calculated by summing all activities which were sufficient to raise breathing rate, as follows:
  (Days of walking * usual minutes of walking IF sufficient to raise breathing rate) + (Days of cycling * usual munities of cycling IF sufficient to raise breathing rate) + (days of sport, fitness or dance * usual minutes of sport, fitness or dance IF sufficient to raise breathing rate).

SECONDARY OUTCOMES:
Cost savings to health care service | 12 months
  Extrapolating the potential cost savings to the health care service of the community programme by analysing the biomarker trend information

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Bottoms, PhD, Principal Investigator — University of Hertfordshire; Daniel Grant, MBBS, Principal Investigator — Medichecks
Locations (1):
- University of Hertforshire, Hatfield, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised group data will be available.

DOCUMENTS (1):
  • Informed Consent Form (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT03809871/ICF_000.pdf